CLINICAL TRIAL: NCT06170801
Title: Efficacy and Feasibility of a Transdiagnostic Augmentation Therapy for Improving Interpersonal Skills Using the Kiesler Circle Training (KCT)
Brief Title: Group Intervention for Interpersonal Skills
Acronym: GRIPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other); University of Greifswald (Other)
Responsible Party: Principal Investigator, Anne Guhn, Dr. rer. nat., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 457376358
Record Dates: First submitted 2023-12-04; First posted 2023-12-14 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Depressive Disorder; Anxiety Disorder
Keywords: Psychotherapy; Depression; Anxiety; Outpatient Treatment; Group Therapy; Childhood Maltreatment; Moderator; Mediator; Daily Social Contacts; Electronical Momentary Assessment; Efficacy; Feasibility
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: prospective, bicenter, evaluator- and statistician-blinded, randomized clinical trial with an active control condition
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of interventions, blinding of patients/therapists concerning the treatment is impossible, but all assessments as well as data analysis will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kiesler Circle Training (KCT) + Cognitive Behavioral Therapy (CBT) (Experimental): The Kiesler Circle Training (KCT) consists of 12 weekly group sessions of 100 minutes each (in a group of max. 10 patients). In addition, all patients receive weekly individual state-of-the-art CBT sessions (50 minutes each).
  Interventions: Behavioral: Kiesler Circle Training (KCT); Behavioral: Cognitive Behavioral Therapy (CBT)
- Cognitive Behavioral Therapy (CBT) (Active Comparator): The patients receive weekly individual state-of-the-art CBT sessions (50 minutes each).
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Kiesler Circle Training (KCT) — Kiesler Circle Training is a transdiagnostic modular group treatment, which comprises a baseline module and four additional independent modules (nonverbal communication, verbal communication, conflict training and empathy and corrective interpersonal experiences). KCT is based on a heuristic model to explain and anticipate interactions developed by Donald Kiesler and other representatives of the interpersonal theory. The circumplex model arranges the variety of interpersonal behaviors in terms of a circular continuum allocated on two orthogonal axes: The vertical axis addresses interpersonal control (agency), the horizontal axis addresses interpersonal communion. The model further allows illustrating complementary action tendencies to anticipate other's reactions and to guide own behavior to achieve interpersonal goals. KCT is designed for increasing the awareness of such interpersonal action tendencies and for improving interpersonal behavioral flexibility.
  Arms: Kiesler Circle Training (KCT) + Cognitive Behavioral Therapy (CBT)
Behavioral: Cognitive Behavioral Therapy (CBT) — Cognitive Behavioral Therapy is based on the interrelationships of thoughts, actions and feelings. Presumably, individual CBT will address intrapersonal therapeutic foci such as behavioral activation, identification of dysfunctional thoughts, overcoming fears by exposure, etc. Individual CBT may also include interpersonal functioning as therapeutic foci. Disorder-specific treatment manuals are available for all diagnoses included in the study. Of note, state-of-the-art CBT does not necessarily mean, that individual CBT-sessions strictly adhere to a manual. However, because both study sites are CBT training institutes, which guarantee supervision at least every four hours, it can be estimated that state-of-the-art CBT is realized.

SUMMARY:
The purpose of this study is to compare an individual state-of-the-art cognitive behavioral therapy (CBT) with CBT augmented by a group intervention for improving interpersonal skills, the Kiesler Circle Training (CBT+KCT), in patients with a depressive or anxiety disorder.

DETAILED DESCRIPTION:
This study aims to test the effectiveness and feasibility of a transdiagnostic group psychotherapy to improve interpersonal skills, the Kiesler Circle Training (KCT). For this purpose, a prospective, bicentre, randomised clinical trial (RCT) blinded by evaluators and statisticians will be conducted on outpatients with diagnoses of anxiety and/or depressive disorders according to DSM-5. An individual state-of-the-art cognitive behavioral therapy (CBT) will be compared with CBT augmented by Kiesler Circle Training (CBT + KCT) in a sample of 156 patients (CBT: 78 patients, CBT + KCT: 78 patients). All participants will be assessed four times, at baseline (T1, week 2), at mid-treatment (T2, week 9), at post-treatment (T3, week 14) and at 3-months follow-up (T4, week 26). Outcome measurements include interpersonal problems as well as symptom change in regard to both the categorical approach (primary diagnosis) and the transdiagnostic approach. The two main hypotheses are:

1. the improvement of interpersonal problems in the experimental group (CBT + KCT) will be greater than the improvement in the control group (CBT).
2. the improvement of interpersonal problems will be associated with decreasing symptom severity related to the primary diagnosis, so that patients in the conjoint CBT+KCT treatment will reach higher symptom change scores than patients in the CBT only condition.

Furthermore, we assume that the course of interpersonal problems is moderated by childhood maltreatment and mediated by the quality and quantity of daily social contacts.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient knowledge of the German language (B2 level)
* Primary diagnosis of either depressive disorder or anxiety disorder according to DSM-5 at time of screening
* Interpersonal distress above average (IIP-32 > 1.81) at time of screening
* Ongoing individual CBT at time of screening
* Signed informed consent regarding the study protocol

Exclusion Criteria:

* Acute suicidality at time of screening
* Active substance abuse at time of screening
* Borderline, antisocial, schizoid or schizotypic personality disorder at time of screening
* Inability to participate in outpatient treatment with additional weekly group appointment at time of screening
* Any kind of additional group treatment (including self-help groups) besides individual CBT during the entire study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Inventory for Interpersonal Problems (IIP-32; Horowitz et al., 1988, German: Thomas et al., 2011) | Weeks 1, 14
  Change in interpersonal functioning, measured with the IIP-32 from baseline (Time 1) to week 14 (Time 2), represents the primary outcome measure. The IIP-32 is a self-assessment questionnaire for interpersonal problems, i.e., difficulties in interacting with other individuals, based on Horowitz's Circumplex Model. It consists of 32 items that are answered on a 5-point scale (0= not at all, 4 = very much). For evaluation, a mean score is calculated across all items, with a higher score indicating a higher severity of interpersonal problems.

SECONDARY OUTCOMES:
Inventory for Interpersonal Problems (IIP-32; Horowitz et al., 1988, German: Thomas et al., 2011) | Baseline, Weeks 1, 9, 14, 26
  The IIP-32 is a self-assessment questionnaire for interpersonal problems, i.e., difficulties in interacting with other individuals, based on Horowitz's Circumplex Model. It consists of 32 items that are answered on a 5-point scale (0= not at all, 4 = very much). For evaluation, a mean score is calculated across all items, with a higher score indicating a higher severity of interpersonal problems.
Impact Message Inventory, revised version (IMI-R; Kiesler et al., 2006; German: Caspar et al., 2016) | Weeks 1, 14, 26
  As key secondary endpoint, observer-rated changes in interpersonal functioning from Time 1 (week 1) to Time 2 (week 14) will be investigated with the IMI-R. The IMI-R will be conducted by blinded study raters. The IMI-R uses 64 items (8 items for each Kiesler Circle position) to capture covert reactions that a patient evokes in a blinded-rater. Through this assessment, it is possible to create an individual Kiesler Circle profile for each patient. The assessment of each behavior is conducted on a 4-point scale (1 = strongly disagree; 4 = strongly agree), so that higher values mean a higher expression of the Kiesler Circle position.
Hamilton Depression Rating Scale, 24 items version (HAM-D, Hamilton, 1967) | Weeks 1, 9, 14, 26
  The HAMD is a semi-structured interview, which measures the severity of depressive symptoms experienced in the last week. Blinded study raters will assess the severity of symptoms for each of the 24 items using a scale ranging from 0-2, 0-3, or 0-4. The total score ranges from 0-75, with higher scores indicating a higher severity of depression.
Beck Depression Inventory, simplified (BDI-V; Beck, 1961; German version: Schmitt et al., 2000) | Weeks 1, 9, 14, 26
  The BDI-V is a self-report questionnaire designed to assess the severity of depressive symptoms. Patients rate the severity of 20 depression symptoms on a 6-point scale (0 = never, 5 = almost always). The total score ranges from 0 to 100, with higher scores indicating a higher severity of depression.
Hamilton Anxiety Rating Scale (HAM-A; Hamilton, 1959) | Weeks 1, 9, 14, 26
  The HAM-A is a clinician-rating to assess the severity of anxiety symptoms experienced in the last week. Blinded raters will assess the severity of symptoms for each of 14 items using a 5-point scale ranging from 0 to 4. The total score ranges from 0 to 56, with higher scores indicating a higher severity of anxiety.
Questionnaire on panic-related Anxieties, Cognitions and Avoidance (ACA; Chambless et al., 1984; German: Ehlers et al., 2001) | Weeks 1, 9, 14, 26
  The ACA is a self-report questionnaire of which we assess two subdomains in our study: the Body Sensations Questionnaire (BSQ) and the Agoraphobic Cognitions Questionnaire (ACQ). The BSQ asks about anxiety regarding 17 physical symptoms and the ACQ about 14 catastrophizing thoughts that can occur during anxiety. Answers are given on a 5-point scale, with higher scores indicating higher levels of anxiety (1 = not anxious/never, 5 = extremely anxious/always). A mean value is calculated for each of the two subdomains.
Short Emotional Disorder Inventory (SEDI; adopted short version of the MEDI by Kaiser et al., unsubmitted) | Weeks 1, 14, 26
  The SEDI is a short form of the Multidimensional Emotional Disorder Inventory (MEDI; Rosellini & Brown, 2019), which represents a dimensional approach to classify emotional disorders. The SEDI is a self-report questionnaire comprising 15 items that are answered on a 4-point scale (1 = completely untrue or slightly true, 4 = completely true). A mean value is calculated over all items, with higher values indicating a higher level of emotional disorder traits.
Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001) | Weeks 1, 14, 26
  The PHQ-9 is part of the Patient Health Questionnaire and measures depressive symptoms using 9 items. The rating scale is 4-point (0 = never, 3 = almost daily) and a total score ranging from 0-24 is calculated.
Patient Health Questionnaire-15 (PHQ-15; Kroenke et al., 2002) | Weeks 1, 14, 26
  The PHQ-15 is part of the Patient Health Questionnaire and measures the 15 most common somatic symptoms of outpatients. The rating scale is 3-point (0 = not affected, 2 = severely affected) and a total score ranging from 0-30 is calculated.
Generalized Anxiety Disorder 7 (GAD-7; Spitzer et al., 2006) | Weeks 1, 14, 26
  The GAD-7 was integrated into the patient health questionnaire in 2006 as a validated scale for measuring generalized anxiety disorder using 7 items. The rating scale is 4-point (0 = never, 3 = almost daily) and a total score ranging from 0-21 is calculated.
World Health Organization Quality of Life (WHOQoL-BREF; The WHOQOL Group, 1998) | Weeks 1, 14, 26
  The WHOQoL-BREF is a self-report measure and assesses the subjective quality of life across physical, psychological, social, and environmental domains using 26 items. These domains are rated by patients on a 5-point scale and a mean score for each domain is calculated by multiplying the mean value of all items of the respective domain by four. The possible values for all domain scores therefore range from 4-20.
Personality Inventory for DSM-5 Brief Form Plus (PID5BF+M; Bach et al., 2020) | Weeks 1, 14, 26
  The PID5BF+M is a self-report questionnaire designed to assess maladaptive personality traits in alignment with the DSM-5 and ICD-11. The questionnaire comprises 36 items, which are answered on a 4-point scale (0 = completely untrue, 3 = completely true) and captures six personality trait domains (negative affectivity, detachment, antagonism/dissociality, disinhibition, anankastia, and psychoticism). A mean value is calculated for each domain, with higher scores indicating higher expression of that personality domain.
Level of Personality Functioning Scale-Brief Form 2.0 (LPFS-BF; Spitzer et al., 2021) | Weeks 1, 14, 26
  The LPFS-BF is a self-report questionnaire designed to assess personality functioning in alignment with the DSM-5 and ICD-11. The questionnaire comprises 12 items, which are answered on a 4-point scale (1 = completely untrue, 4 = completely true) and captures two personality functioning domains (self and interpersonal pathology). A mean value is calculated for each domain, with higher scores indicating higher expression of that personality functioning domain.
Interpersonal Needs Questionnaire (INQ; Forkmann, T. & Glaesmer, H., 2013) | Weeks 1, 14, 26
  The Interpersonal Needs Questionnaire (INQ) measures interpersonal needs using two subscales: thwarted belongingness and perceived burdensomeness. The questionnaire consists of 15 items, that are answered on a 7-point scale (1 = completely untrue, 7 = completely true). After reversing the polarity of 6 items, a mean value is calculated for each of the two subscales, with higher scores indicating higher levels of thwarted belongingness and perceived burdensomeness.

OTHER OUTCOMES:
Childhood Trauma Questionnaire (CTQ; Original: Bernstein & Fink, 1998; German: Wingenfeld et al., 2010) | Baseline
  Childhood maltreatment is assessed as a main moderator at baseline. The CTQ is a self-report assessment designed to measure experiences of childhood trauma and abuse on five subscales (emotional abuse, physical abuse, sexual abuse, emotional neglect and physical neglect). Patients rate the frequency of 34 of these experiences on a 5-point scale (1= not at all, 5 = very often), and each subscale score has a range from 5 to 25 points. Higher scores indicate a higher severity in childhood trauma.
Quality and quantity of daily social contacts | Three one-week EMA surveys (3 weeks in total: week 1-2, week 8-9, week 15-16)
  Patients answer short questionnaires four times a day, which appear on their smartphone at random times (Electronical Momentary Assessment, EMA). The number of social contacts, the quality of social contacts (interpersonal complementarity), interaction partner, affect and anxiety are assessed.
Inventory for the Assessment of Negative Effects of Psychotherapy (INEP; Ladwig et al., 2014) | Weeks 1, 14, 26
  The INEP is a self-report assessment of negative changes caused by psychotherapy in the areas of intrapersonal change, relationships, friendships, family, malpractice, and stigmatization. The INEP contains 21 items, which responses are partly formulated in a 7-point bipolar format (-3 = negative change is completely true, 0 = unchanged, 3 = positive change is completely true), and partly formulated in a 4-point unipolar format (0 = completely untrue; 3 = completely true). In addition, patients' attributions regarding the cause of negative effects is assessed. For the evaluation, only negative effects directly attributed to the psychotherapeutic treatment are considered.
Questionnaire for the Assessment of Side Effects and Negative Experiences in Group Therapy (NUGE- 24; Strauß & Drobinskaya, 2018) | Weekly during the weeks 3-14
  The NUGE assesses adverse experiences with group psychotherapy and side effects of the group setting by differentiating between group-related and therapist-related stress, stress from co-patients and personal overload. The NUGE comprises 24 items and responses are given on a 5-point scale (1 = strongly disagree, 5 = strongly agree), with higher scores indicating higher distress. The NUGE will be completed after each KCT group session by patients randomly assigned to the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Guhn, Dr., Principal Investigator — Charite University, Berlin, Germany; Eva-Lotta Brakemeier, Prof. Dr., Principal Investigator — University of Greifswald
Locations (1):
- Charité, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Following the Open Science guidelines of the German Psychological Association (DGPS), anonymized data will be made available via the Open Data portal of the Open Science Foundation (www.osf.io). The data will be stored after the completion of data collection, but not before 01.06.2026. This practice enables external parties to replicate the analyses mentioned in scientific publications and to perform ad hoc analyses. The data is permanently stored on servers located in Germany. Once uploaded and published, these anonymized data cannot be deleted and are exempt from deletion even if a study participant later decides to revoke their participation.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: We will make the outcome data and then the covariate data freely available after our respective publications, but not before 01.06.2026.
Access Criteria: Data will be shared with the public; data will be made available for all what types of analyses; the mechanism by which the data will be made available will be determined soon.

REFERENCES:
- [Derived] Ollrogge K, Schulze D, Sterzer P, Kohler S, Friedel E, Romanczuk-Seiferth N, Siegerist AL, Brakemeier EL, Guhn A. Cognitive behavioural therapy plus Kiesler Circle Training (CBT+) versus CBT only for patients with interpersonal problems: study protocol for a randomised controlled feasibility trial. BMJ Open. 2025 Feb 11;15(2):e098466. doi: 10.1136/bmjopen-2024-098466. PMID 39933819